CLINICAL TRIAL: NCT07117448
Title: Relationship Between Clinical and Radiological Parameters, Static and Dynamic Balance, Pain, Quality of Life and Body Image in Adolescents With Scheuermann's Kyphosis
Brief Title: Clinical and Radiological Correlates of Balance, Pain and Body Image in Adolescents With Scheuermann's Kyphosis
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sılanur Güney Çamlıca, Medical Doctor, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: 24/543
Record Dates: First submitted 2025-06-18; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Scheuermann Disease
Keywords: Kyphosis; Balance; Sagittal balance; Spinopelvic parameters; Scheuermann Disease
MeSH Terms: conditions — Scheuermann Disease; Kyphosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Scheuermann's Kyphosis Group: Adolescents diagnosed with Scheuermann's kyphosis according to Sorensen criteria
- Healthy Control Group: Age- and sex-matched healthy adolescents with no spinal deformity

SUMMARY:
The goal of this observational study is to evaluate the relationship between sagittal and spinopelvic radiological parameters of the spine and clinical outcomes in adolescents with Scheuermann's kyphosis (SK) by assessing dynamic and static balance, pain, quality of life, and body image. The main questions it aims to answer are: Is there a correlation between kyphosis severity, spinopelvic measurements, and balance scores in adolescents with Scheuermann's kyphosis? How do pain, body image, and quality of life relate to radiological parameters and clinical findings in these individuals? Are there significant differences in balance, spinopelvic parameters, body image, and quality of life between adolescents with Scheuermann's kyphosis and healthy controls?

Participants will undergo radiological evaluation of sagittal spine and spinopelvic parameters using standing lateral spinal radiographs, static and dynamic balance assessments to evaluate postural stability, pain assessment using validated pain scales, and quality of life and body image assessments through standardized questionnaires.

Researchers will compare Scheuermann's kyphosis patients and age-matched healthy controls to determine the impact of kyphosis severity on balance, body image, and quality of life.

DETAILED DESCRIPTION:
Scheuermann's disease, also known as juvenile kyphosis or juvenile discogenic disease, is a hyperkyphotic condition of the spine involving the vertebral bodies and discs, defined by anterior wedging of 5 degrees or more in three or more consecutive vertebral bodies. Some studies suggest that a single wedged vertebra associated with irregular vertebral endplates is sufficient for diagnosis. The thoracic spine is most commonly affected, but involvement may also extend to the thoracolumbar/lumbar region. The estimated prevalence in the general population is 0.4-8%, with a similar male-to-female ratio.

The exact and universally accepted etiology of Scheuermann's kyphosis (SK) has yet to be determined. It is suggested that disproportionate vertebral endplate mineralization and ossification during growth lead to uneven vertebral body growth, ultimately resulting in kyphosis with the characteristic wedge-shaped vertebral bodies. Thoracic hyperkyphosis in individuals with flexible spines is typically compensated by non-structural hyperlordosis of the lumbar and cervical spine. The head and shoulders are positioned forward, and the deformity is relatively fixed, not resolving with hyperextension. Neurological examination is almost always normal. The diagnosis is often made in adolescents aged 12 to 17 years when parents notice a postural deformity or hunchback appearance. Pain in the affected hyperkyphotic region may be the reason for initial evaluation, which may worsen with standing and activity but typically resolves upon skeletal maturity. The extent and severity of pain vary based on the patient's age, disease stage, kyphosis location, and deformity severity. In addition to spinal deformity, these patients often experience tightness in the pectoral, hamstring, and iliopsoas muscles.

For imaging, standard standing lateral and anteroposterior spinal radiographs are essential. The kyphosis angle is measured on lateral radiographs using the Cobb method. The normal range of thoracic kyphosis, according to the Scoliosis Research Society (SRS), is 20°-40° using the Cobb method. Based on the apex of kyphosis, SK is classified as thoracic type if the apex is at T7-T9, thoracolumbar type if at T10-T12, and lumbar type in cases with progressive low back pain, decreased lumbar lordosis, and characteristic radiographic changes.

The importance of sagittal profile assessment in spinal pathologies is increasing. Neutral sagittal balance is evaluated on standing lateral spinal radiographs. Kyphotic deformities disrupt neutral sagittal balance. Increased kyphotic deformity causes the head to shift forward beyond the feet and pelvis, resulting in positive sagittal imbalance.

Balance includes static balance, which is the ability to maintain the body in a specific position; dynamic balance, which is the ability to maintain balance during movement; and postural stability, which is the ability to maintain orientation in relation to the surrounding environment. This mechanism involves a neuromuscular interaction that integrates information from proprioceptive, visual, and vestibular inputs to generate an appropriate motor response to keep the body's center of mass within the base of support. Morphological spinal deformities can alter head position, lead to asymmetric muscle activity around the spine, and shift the body's center of mass, affecting postural stability and balance performance. Therefore, postural stability and balance performance in upright standing may be altered in individuals with spinal deformities such as scoliosis and hyperkyphosis. A kyphotic posture may cause the center of mass to shift forward beyond stability limits, reducing postural balance and increasing fall risk. Dysfunction in somatosensory pathways may impair postural control mechanisms, potentially influencing the etiology or progression of scoliosis.

The literature associates different scoliotic curvatures with altered posturography and postural sway under both static and dynamic conditions, indicating varying degrees of balance impairment. Some studies suggest that the degree of balance dysfunction correlates with the severity of the scoliotic curvature. While previous studies on SK have examined the relationship between radiographic findings and clinical symptoms, the impact of abnormal thoracic kyphotic posture on static balance, and spinopelvic parameters between SK patients and age-matched controls, no study has compared kyphosis severity and spinopelvic measurements with balance scores, body image, and quality of life.

This study aims to investigate the relationship between sagittal and spinopelvic radiological parameters and clinical findings in adolescents with Scheuermann's kyphosis by evaluating dynamic and static balance, pain, quality of life, and body image. Additionally, changes in these parameters will be compared with those of healthy adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 10 to 18 years
* Diagnosis of Scheuermann's kyphosis based on Sorensen criteria (for patient group)
* Healthy volunteers matched for age and sex (for control group)
* Ability to understand and comply with study procedures
* Informed consent obtained from participants and/or guardians

Exclusion Criteria:

* Neuromuscular disorders
* History of spinal surgery or traumatic spinal injury
* Scoliosis > 15° (Cobb angle)
* Vestibular, visual, or auditory impairments
* Lower extremity musculoskeletal disorders affecting gait or balance
* Cognitive or psychiatric conditions affecting participation
* Use of orthotic devices or braces
* Any other systemic condition affecting postural control

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents aged 10 to 18 years, including individuals diagnosed with Scheuermann's kyphosis and age- and sex-matched healthy controls. All participants were recruited from the department of physical medicine and rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Balance Parameters Assessed by Multiple Modalities | At enrollment (Day 0, cross-sectional)
  Clinical balance tests will assess static postural control by recording the duration (in seconds) the participant maintains the test position.
  Stabilometric platform will measure postural sway parameters during quiet stance. Computerized Dynamic Posturography (CDP) will provide composite scores reflecting balance performance under various sensory conditions Each method will be analyzed and reported separately. Additionally, agreement and correlation between clinical balance tests and device-based measurements (stabilometric platform and CDP) will be evaluated.

SECONDARY OUTCOMES:
Pain Level Assessed by Numeric Rating Scale (NRS) | At enrollment (Day 0)
  Pain intensity will be assessed using the Numeric Rating Scale (NRS), ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate greater pain severity.
Health-Related Quality of Life Assessed by SRS-22r | At enrollment (Day 0)
  Quality of life will be evaluated using the SRS-22r questionnaire, consisting of 22 items covering five domains: function, pain, self-image, mental health, and satisfaction. Each item is scored from 1 to 5. Higher scores indicate better quality of life.
Body Image Perception Assessed by SAAS | At enrollment (Day 0)
  Body image perception will be evaluated using the Social Appearance Anxiety Scale (SAAS), a 16-item self-report scale. Items are scored on a 5-point Likert scale from 1 (not at all) to 5 (extremely). Higher scores reflect greater appearance-related anxiety and more negative body image.
Correlation Between Clinical and Radiological Parameters | At enrollment (Day 0)
  Correlations will be analyzed between clinical outcome measures (pain via NRS, quality of life via SRS-22r, and body image via SAAS) and radiographic parameters (e.g., kyphosis angle, pelvic incidence, sagittal vertical axis). Statistical analyses will include correlation coefficients to assess the strength and direction of associations.

CONTACTS AND LOCATIONS:
Overall Officials: sılanur güney çamlıca, medical doctor, Principal Investigator — Resident University of Health Sciences, FSM Training and Research Hospital, Istanbul
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided